CLINICAL TRIAL: NCT02532608
Title: Infra-slow Oscillations During Sleep, After Acute Sleep Deprivation and in Subjects With Restless Legs Syndrome/Periodic Leg Movements During Sleep (RLS/PLMS): an Explorative, Prospective, Monocentric, Observational Case-control and Interventional Study
Brief Title: Infra-slow Oscillations During Sleep
Acronym: SleepD-ISO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stephany Fulda (Other)
Responsible Party: Sponsor-Investigator, Stephany Fulda, PhD, Neurocenter of Southern Switzerland
Organization: Neurocenter of Southern Switzerland (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EOC.NSI.LS.15.2
Record Dates: First submitted 2015-08-21; First posted 2015-08-26 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Healthy Subjects; Restless Legs Syndrome; Periodic Limb Movements During Sleep
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acute sleep deprivation (Experimental): Registration of habitual sleep and sleep after sleep deprivation
  Interventions: Other: Acute sleep deprivation

INTERVENTIONS:
Other: Acute sleep deprivation — Participants will stay awake for 36 hours

SUMMARY:
In this study the investigators plan to systematically characterise infra-slow EEG oscillations during sleep, explore their relationship to the microstructure of sleep, and investigate its role in the physiology and pathophysiology of sleep by co-registration of Full band EEG with polysomnography during wake and sleep in healthy subjects, after sleep deprivation, and in patients with restless legs syndrome/periodic leg movements during sleep (RLS/PLMS).

DETAILED DESCRIPTION:
Sleep is a highly dynamic process and during large parts of sleep the level of arousal fluctuates on a multi-second time scale between the sleep stage specific background and transient, phasic events that clearly arise from this background and constitute the microstructure of sleep. This microstructure is part of the dynamic physiological sleep regulation and at the same time reflects the instability of sleep, is critically involved in the pathophysiology of sleep and a determinant of the recuperative value of sleep and daytime performance.

Intriguingly, these sleep microstructural fluctuations are in a multi-second range that corresponds closely to the so-called infra-slow oscillations that are ubiquitous in the central nervous system. Infra-slow oscillations (0.01 - 0.1 Hz) have been observed in both humans and animals across brain structures and spatial scales in the dynamics of single unit firing rates, direct electrical potential fluctuations and oscillation amplitude modulations. The possibility to record these infra-slow oscillations on the level of the surface EEG with direct current (DC) or Full band (Fb) EEG offers a new approach to study the microstructure of sleep and characterise the full range of sleep-related EEG oscillations.

The objectives of this study are:

1. to record and systematically characterise infra-slow oscillations during wake and all stages of sleep
2. to explore the relationship between sleep infra-slow oscillations and microstructural events of sleep, in particular the cyclic alternating pattern
3. to explore the effect of acute sleep deprivation on sleep infra-slow EEG activity
4. to investigate infra-slow sleep EEG activity in patients with RLS/PLMS, common sleep disorders with prominent periodic arousals, heart rate activations, and leg movements
5. to explore the relationship between infra-slow EEG oscillations and periodic events in movement and autonomic system activity in patients with RLS/PLMS.

ELIGIBILITY:
Inclusion Criteria for all participants:

* Willingness to participate and written informed consent
* Aged 20 to 40 years at the time of screening
* Body mass index (BMI) ≤ 30

Additional inclusion criteria for subjects with RLS/PLMS:

* Either diagnosis of RLS and current IRLS score ≥ 15.
* Or frequent periodic leg movements during sleep

Exclusion criteria for all participants:

* Pregnancy or breast feeding at the time of screening
* Sleep related breathing disorders
* Current psychiatric disorders
* Current chronic treatment that may affect sleep.
* Any significant neurological disorder or other medical disease that may affect sleep.
* Any unstable medical condition.

Additional exclusion criteria for participants with RLS/PLMS:

* Current intake of dopaminergic drugs
* Current intake of other RLS relevant medication
* Intake of hypnotics
* Other significant sleep disorder except symptoms potentially related to RLS

Additional exclusion criteria for healthy participants:

* Any pharmacological treatment that may affect sleep and/or sleep related movement disorders
* Any clinically significant sleep disorders

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-10; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Infra-slow frequency power | 36 hours
  Average power (µV) in the infra-slow frequency range during wake and different stages of sleep derived from standard fast fourier transform and continuous wavelet transform.

CONTACTS AND LOCATIONS:
Overall Officials: Stephany Fulda, PhD, Principal Investigator — Neurocenter of Southern Switzerland
Locations (1):
- Neurocenter of Southern Switzerland, Lugano, Canton Ticino, Switzerland